CLINICAL TRIAL: NCT06908408
Title: Correlation Between the Severity of Metabolic Acidosis in Patients on Admission to the ICU and Platelet Count Trend in the Following Days
Brief Title: Correlation Between Base Excess in Patients Upon Admission to the ICU and Platelet Count Trend in the Following Days
Acronym: BE-Platelet
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Irena Grad, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: UMCLj-BE-Platelet; Irena Grad (Other: UMCLjubljana)
Record Dates: First submitted 2025-03-22; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Platelet Count Decline in Critically Ill; Metabolic Acidosis; Metabolic Acidosis Severity; Platelet Count Decline in ICU Patients
Keywords: metabolic acidosis severity; BE; relative platelet count decline in critically ill; base excess; platelet count decline in critically ill
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Corrrelation between metabolic acidosis severity in patients on admission to the ICU and platelet count trend in 2 days following admission was investigated — The aim of the study was to investigate if there exists any correlation between metabolic acidosis severity in patients upon admission to the ICU and platelet count trend in 2 days, following admission.

SUMMARY:
Several studies have revealed that a relative platelet count decline in patients after their admission to the intensive care unit (ICU) is a very reliable marker of the severity of their sickness. ICU patients with a greater platelet count decline after their admission to the ICU have generally worse outcome. Investigators assume that a quick appearance of a deep metabolic acidosis, which commonly occurs in critically ill, has an important role in pathogenesis of relative platelet count decline. To evaluate this, correlation of metabolic acidosis severity in participants upon admission to the ICU with platelet count decline in 2 days, following admission, was investigated with a retrospective observational study, analysing all participants, admitted to the ICU in one year period (in 2020).

As a measurement of metabolic acidosis severity, investigators took base excess (BE) value (expressed in mmol/L) from arterial blood gas analysis with lowest pH in participants in around admission time (in a period from 24 hours before to 24 hours after their admission to the ICU). To calculate relative platelet count decline in 2 days after admission to the ICU, investigators took platelet count on admission to the ICU (P0) and lowest platelet count on day 2 after the patient's admission (P2). Following formula was used to calculate relative platelet count decline in 2 days after ICU admission (delta P): delta P = (P2-P0)/P0 x 100 (expressed in %). More negative values of delta P represent larger relative platelet count decline.

The main interest of the study was if BE value correlates with delta P. Investigators assumed that participants with a more severe metabolic acidosis upon admission to the ICU (represented with more negative BE value) would tend to have a larger relative platelet count decline in 2 days, following admission to the ICU (represented with more negative value of delta P).

Pearson correlation was used to evaluate correlation between BE and delta P.

DETAILED DESCRIPTION:
The aim of the study was to answer the question, if metabolic acidosis severity in participants upon admission to the ICU correlatets with platelet count decline in days, following admission.

Investigators conducted this study at the Department of Anesthesiology and Surgical Intensive Care at University Medical Centre Ljubljana. The study included all participants, admitted to the ICU in a one-year period (in 2020; from 1st January to 31st December 2020). From the electronic recordings of the department (Hospital Information System BIRPIS21), investigators obtained the following data of each participant: age, gender, lowest pH in arterial blood gas analysis in around admission time with corresponding bicarbonate concentration [HCO3-] and BE value, platelet count on admission (P0), and lowest platelet count on second day after ICU admission (P2).

As a measurement of metabolic acidosis severity, investigators took the BE value of arterial blood gas analysis with the lowest pH from the range of 24 hours before to 24 hours after ICU admission. To calculate relative platelet count decline in 2 days after ICU admission (delta P), the following formula was used: delta P = (P2-P0)/P0 x 100.

Participants who died before the second day after ICU admission or participants whose demanded laboratory findings were for some other reasons lacking (arterial blood gas analysis or platelet count on admission or platelet count on second day after ICU admission), were excluded from final analysis of correlation between BE and delta P.

Pearson's correlation coefficient (r) with 95% confidence interval (CI) was used to estimate the association between BE and delta P.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU department in a 1 year period (from 1st January to 31th December 2020)

Exclusion Criteria:

* Lacking blood gas analysis data on admission
* Incomplete platelet count data (lacking platelet count on admission to the ICU and day 2 after the admission)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study has been conducted at the Department of Anaesthesiology and Surgical Intensive Care at University Medical Centre Ljubljana. All participants, admitted to the ICU of Department of Anaesthesiology and Surgical Intensive Care in 2020 were included.
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Relative platelet count decline in participants from admission to the ICU to their second day after ICU admission | From admission to the ICU (base line) and 2 days following admission
  In this observational study relative platelet count decline in participants from admission to the ICU to their second day after the admission to the ICU was measured (with the aim to analyse correlation between metabolic acidosis severity in participants upon admission to the ICU and platelet count trend in participants in the following 2 days).
  Platelet count value in participants upon admission to the ICU (P0) and lowest platelet count value on day 2 after the admission to the ICU (P2) were used to calculate relative platelet count decline in 2 days after ICU admission (delta P), using formula: delta P = (P2-P0)/P0 x 100 (delta P expressed in %).

CONTACTS AND LOCATIONS:
Overall Officials: Primož Gradišek, MD, PhD, Prof., Study Chair — Department of Anaesthesiology and Surgical Intensive Care
Locations (1):
- University Medical Centre Ljubljana, Zaloška cesta 7, 1000 Ljubljana, Slovenia, Ljubljana, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning with publication of results with no end date.
Access Criteria: After publication of results all IPD data of the study can be shared on request on email of investigator: irena.grad@gmail.com

REFERENCES:
- [Background] Patel JK, Kataya A, Parikh PB. Association between intra- and post-arrest hyperoxia on mortality in adults with cardiac arrest: A systematic review and meta-analysis. Resuscitation. 2018 Jun;127:83-88. doi: 10.1016/j.resuscitation.2018.04.008. Epub 2018 Apr 10. PMID 29653154
- [Background] Demiselle J, Wepler M, Hartmann C, Radermacher P, Schortgen F, Meziani F, Singer M, Seegers V, Asfar P; HYPER2S investigators. Hyperoxia toxicity in septic shock patients according to the Sepsis-3 criteria: a post hoc analysis of the HYPER2S trial. Ann Intensive Care. 2018 Sep 17;8(1):90. doi: 10.1186/s13613-018-0435-1. PMID 30225670
- [Background] Roberts BW, Kilgannon JH, Hunter BR, Puskarich MA, Pierce L, Donnino M, Leary M, Kline JA, Jones AE, Shapiro NI, Abella BS, Trzeciak S. Association Between Early Hyperoxia Exposure After Resuscitation From Cardiac Arrest and Neurological Disability: Prospective Multicenter Protocol-Directed Cohort Study. Circulation. 2018 May 15;137(20):2114-2124. doi: 10.1161/CIRCULATIONAHA.117.032054. Epub 2018 Feb 1. PMID 29437118
- [Background] Geers C, Gros G. Carbon dioxide transport and carbonic anhydrase in blood and muscle. Physiol Rev. 2000 Apr;80(2):681-715. doi: 10.1152/physrev.2000.80.2.681. PMID 10747205
- [Background] Park MAJ, Cave G, Freebairn RC. Metabolic acidosis in anaesthesia and critical care. BJA Educ. 2024 Mar;24(3):91-99. doi: 10.1016/j.bjae.2023.12.005. Epub 2024 Jan 22. No abstract available. PMID 38375495
- [Background] Scardina P, Edwards M. Prediction and measurement of bubble formation in water treatment. Journal of Environmental Engineering 2001 Nov;127:968-973.
- [Background] Pontier JM, Jimenez C, Blatteau JE. Blood platelet count and bubble formation after a dive to 30 msw for 30 min. Aviat Space Environ Med. 2008 Dec;79(12):1096-9. doi: 10.3357/asem.2352.2008. PMID 19070304
- [Background] Pontier JM, Blatteau JE, Vallee N. Blood platelet count and severity of decompression sickness in rats after a provocative dive. Aviat Space Environ Med. 2008 Aug;79(8):761-4. doi: 10.3357/asem.2299.2008. PMID 18717114
- [Background] Levi M, Opal SM. Coagulation abnormalities in critically ill patients. Crit Care. 2006;10(4):222. doi: 10.1186/cc4975. PMID 16879728
- [Background] Ilker Hayiroglu M, Cinar T, Ilker Tekkesin A. Intra-aortic balloon pump-related thrombocytopenia: Its effects on in-hospital mortality in cardiogenic shock patients. Annals Med Res 2021;26(7):1388-93.
- [Background] Vanderschueren S, De Weerdt A, Malbrain M, Vankersschaever D, Frans E, Wilmer A, Bobbaers H. Thrombocytopenia and prognosis in intensive care. Crit Care Med. 2000 Jun;28(6):1871-6. doi: 10.1097/00003246-200006000-00031. PMID 10890635
- [Background] Wang L, Shao J, Shao C, Wang H, Jia M, Hou X. The Relative Early Decrease in Platelet Count Is Associated With Mortality in Post-cardiotomy Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation. Front Med (Lausanne). 2021 Nov 4;8:733946. doi: 10.3389/fmed.2021.733946. eCollection 2021. PMID 34805203
- [Background] Lee HH, Hong SJ, Ahn CM, Yang JH, Gwon HC, Kim JS, Kim BK, Ko YG, Choi D, Hong MK, Jang Y. Clinical Implications of Thrombocytopenia at Cardiogenic Shock Presentation: Data from a Multicenter Registry. Yonsei Med J. 2020 Oct;61(10):851-859. doi: 10.3349/ymj.2020.61.10.851. PMID 32975059
- [Background] Moreau D, Timsit JF, Vesin A, Garrouste-Orgeas M, de Lassence A, Zahar JR, Adrie C, Vincent F, Cohen Y, Schlemmer B, Azoulay E. Platelet count decline: an early prognostic marker in critically ill patients with prolonged ICU stays. Chest. 2007 Jun;131(6):1735-41. doi: 10.1378/chest.06-2233. Epub 2007 May 2. PMID 17475637